CLINICAL TRIAL: NCT04991922
Title: BostonGene-Integrated Genomic Registry Study
Brief Title: BostonGene-Integrated Genomic Registry (BIGR)
Status: Recruiting | Type: Observational
Sponsor: BostonGene (Industry)
Responsible Party: Sponsor
Other Study IDs: BG-001
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Malignancy
Keywords: cancer; precision medicine; WES; RNA-seq; immuno-therapy; genomic; transcriptomic; multiomic
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this project is to develop a comprehensive database of genomic, transcriptomic, molecular, and clinical characteristics of oncology patients to discover, define, and develop genomic and transcriptomic markers to improve future clinical outcomes across cancer types

DETAILED DESCRIPTION:
Immuno- and targeted therapies have shown promising results for many types of cancer (1). However, the effectiveness of these treatments is not optimal for many patients (2). Therefore, further research is needed to discover, define, and develop genomic, transcriptomic, and integrated molecular markers that can improve clinical outcomes across cancer types (3). Unfortunately, current research is restricted by the limited availability of genomic and transcriptomic results linked to clinical outcomes (3). This study will allow for the collection of key clinical data, including longitudinal follow-up, linked with individual genetic and molecular findings in a single comprehensive registry-based databank. Analysis of these data may lead to advances across cancer subtypes through the identification of transcriptomic and genomic associations with therapies.

Clinical and pathological information, including detailed genetic information from a participant's tumor biopsy, will be obtained by the research staff for each participant enrolled in the BIGR Study. Clinical information will include relevant details about the patient's diagnosis and treatment and will be stored in a secure electronic registry database. No extra scans or procedures for this study will be collected as part of this study. Information will be collected regarding a participant's initial diagnosis, treatment, and outcome. To obtain this information, study staff will contact participants or a participant's doctor at regular time intervals for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected or confirmed malignancy
2. Planned comprehensive genomic (> 100 genes) and/or molecular analysis; or genomic and/or molecular data available from prior sequencing
3. Baseline demographics and treatment information available
4. Willingness for future contact by BIRG study personnel to provide information regarding associated cancer outcomes and treatment.
5. Signed informed consent to participate in the study.
6. Living in the United States at the time of enrollment

Exclusion Criteria:

Life expectancy < 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be identified for the BIGR study from a larger group of patients undergoing BostonGene clinical testing (e.g., BostonGene Tumor Portrait TestTM).
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2031-07-01 (Estimated); Study Completion 2036-07-01 (Estimated)

PRIMARY OUTCOMES:
association between major finding and outcome, Descriptive | 5 years
  associations between genomic findings and outcomes of cancer patients who have undergone comprehensive sequencing.

SECONDARY OUTCOMES:
Predictive probability | 5 years
  identify molecular findings associated with therapy.
Clinical trials matching | 5 years
  identify and link registry subjects to future molecular-based clinical research

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Fowler, Principal Investigator — BostonGene
Locations (1):
- BostonGene, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Murciano-Goroff YR, Warner AB, Wolchok JD. The future of cancer immunotherapy: microenvironment-targeting combinations. Cell Res. 2020 Jun;30(6):507-519. doi: 10.1038/s41422-020-0337-2. Epub 2020 May 28. PMID 32467593
- [Background] Sambi M, Bagheri L, Szewczuk MR. Current Challenges in Cancer Immunotherapy: Multimodal Approaches to Improve Efficacy and Patient Response Rates. J Oncol. 2019 Feb 28;2019:4508794. doi: 10.1155/2019/4508794. eCollection 2019. PMID 30941175
- [Background] Olivier M, Asmis R, Hawkins GA, Howard TD, Cox LA. The Need for Multi-Omics Biomarker Signatures in Precision Medicine. Int J Mol Sci. 2019 Sep 26;20(19):4781. doi: 10.3390/ijms20194781. PMID 31561483